CLINICAL TRIAL: NCT05713929
Title: Study of Atelectasis by Electrical Impedance Tomography and the Effects of Different Positions on Their Occurrence, Reversibility and Regional Distribution, During General Anesthesia
Brief Title: Study of Atelectasis by Electrical Impedance Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: B4062022000256
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Gynecologic Surgical Procedures; Urologic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: 1. 1st measurement (T0-SPONT): in spontaneous ventilation.
  2. Induction, intubation and mechanical ventilation for 5 minutes.
  3. 2nd measurement (T1-LYING): after induction.
  4. Trendelenburg 30° and ventilatory constant parameters.
  5. 3rd measurement (T2-TREND): after 5 minutes of Trendelenburg.
  6. Division into 2 groups according to randomization:
     I. Supine position and recruitment manoeuvre. 4th measurement after 5 minutes. (T3-RM) II. Either put in the Anti Trendelenburg position. 4th measurement after 5 minutes. (TREND Q3- REV)
  7. Horizontal supine position and surgical incision.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment maneuver (RM) group 1 (Active Comparator)
  Interventions: Other: Recruitment maneuver (RM)
- Reverse Trend (REV TREND) group 2 (Active Comparator)
  Interventions: Other: Reverse Trend (REV TREND)

INTERVENTIONS:
Other: Recruitment maneuver (RM) — performance of a recruitment maneuver of 30 cm H20 for 30 seconds and measurement of electrical impedance
  Arms: Recruitment maneuver (RM) group 1
Other: Reverse Trend (REV TREND) — Place the patient in the reverse trendelenburg position and measuring the electrical impedance after 5 minutes
  Arms: Reverse Trend (REV TREND) group 2

SUMMARY:
The goal of this interventional study is to learn about the effects of different positions on the occurrence, regional distribution and reversibility of atelectasis by using a PulmoVista 500 monitor (Dräger. 23542 Lübeck), during general anesthesia with mechanical ventilation.

The main questions it aims to answer are:

* The increase in atelectasis after induction of general anesthesia in supine and Trendelenburg position compared with baseline (spontaneous breathing)
* The eventual possibility of reversal of atelectasis caused by general anesthesia and Trendelenburg position by reverse Trendelenburg position and recruitment manœuvre.

Participants will be adult, autonomous and able to express their will, undergoing elective gynecological or urological surgery in the extended Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over eighteen years old;
* Requiring laparoscopic gynecological, urological or digestive surgery;
* Surgery requiring Trendelenburg position and tracheal intubation.

Exclusion Criteria:

* Emergency operation;
* Thoracic surgery;
* Pulmonary, cardiac pathology;
* Pregnant woman;
* BMI > 30;
* Comorbidities defined as an American Society of Anesthesiologists physical condition greater than 2;
* Language barrier;
* Refusal of consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of atelectasis after induction of general anesthesia (Time 1) | from the base measure to time 1 (10 minutes)
  percentage
the percentage of atelectasis after being positioned in the trendelenburg position (Time 2) | from the base measure to time 2 (15 minutes)
  percentage

SECONDARY OUTCOMES:
The eventual possibility of reversal of atelectasis by reverse Trendelenburg position and recruitment maneuver (Time 3) | from the base measure to time 3 (20 minutes)
  percentage

CONTACTS AND LOCATIONS:
Locations (1):
- HUB Hôpital Erasme, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lung Recruitment — https://pubmed.ncbi.nlm.nih.gov/11172579/
- See also: Mechanisms of atelectasis in the perioperative period — https://pubmed.ncbi.nlm.nih.gov/20608554/
- See also: Impedance tomography as a new monitoring technique — https://pubmed.ncbi.nlm.nih.gov/20445445/
- See also: Effect of Positive End Expiratory Pressure on regional ventilation during laparoscopic surgery monitored by electrical impedance tomography — https://pubmed.ncbi.nlm.nih.gov/21658014/